CLINICAL TRIAL: NCT01665248
Title: Comparison of 18-F Sodium Fluoride Uptake in Culprit Plaques Between Acute Coronary Syndrome and Stable Angina
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: CHEOL WHAN LEE, MD, PhD. (Other)
Responsible Party: Sponsor-Investigator, CHEOL WHAN LEE, MD, PhD., MD, PhD, CardioVascular Research Foundation, Korea
Organization: CardioVascular Research Foundation, Korea (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AMCCV2012-03
Record Dates: First submitted 2012-08-13; First posted 2012-08-15 (Estimated); Last update posted 2014-07-28 (Estimated); Status verified 2014-07

CONDITIONS: Coronary Artery Diseases
Keywords: 18-F Sodium Fluoride; Acute coronary syndrome; Stable Angina
MeSH Terms: conditions — Coronary Artery Disease; Acute Coronary Syndrome; Angina, Stable | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- stable angina pectoris or acute coronary syndrome (Other)
  Interventions: Other: 18-F Sodium Fluoride Uptake in Positron emission tomography

INTERVENTIONS:
Other: 18-F Sodium Fluoride Uptake in Positron emission tomography

SUMMARY:
The purpose of this study is to evaluate the correlations between active calcification and vulnerable plaque.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 20
* Acute coronary syndrome or stable angina

Exclusion Criteria:

* Contraindications to the use of heparin, aspirin, clopidogrel, stainless metal, contrast media
* Acute ST segment elevation myocardial infarction within 12hours, heart failure, cardiac shock
* Any serious medical comorbidity such that the subject's life expectancy is less than 24 months
* Ejection fraction less than 30
* Serum creatinine level of 1.5mg/dl and over
* Vasculitis
* Unwillingness or inability to cooperate or to give informed consent

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-08; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Standardized 18F-NaF uptake value within the culprit plaque | At the time of diagnosis

SECONDARY OUTCOMES:
The relationship between 18F-NaF uptake value and calcium scores by Multidetector Computed Tomography | at the time of diagnosis
The relationship between 18F-NaF uptake value and plaque types by Multidetector Computed Tomography | at the time of diagnosis
The relationship between 18F-NaF uptake value and biomarkers | at the time of diagnosis
  hs-CRP, Troponin-I
The relationship between 18F-NaF uptake value and invasive imagings | at the time of diagnosis
  Intravascular ultrasound, Optical coherence tomography

CONTACTS AND LOCATIONS:
Overall Officials: Cheol Whan Lee, MD, PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea